CLINICAL TRIAL: NCT06694740
Title: Effect of Interferon Gamma as a Treatment for Post-aggressive Immunosuppression in Intensive Care Units, a Randomized Bayesian Double-blind Controlled Trial Versus Placebo
Acronym: INFINITY
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APHP220672; 2023-506725-11-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-12; First posted 2024-11-19 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Post-aggressive Immunosuppression; Adult Patients Admitted to Intensive Care With Initial Severity (SOFA of the First 24 Hours Post-admission ≥ 6; Adult Under Mechanical Ventilation, and Presenting an mHLA-DR Less Than 8,000AB/C
Keywords: Critical care; ICU-acquired immune suppression; HLA-DR; immunity; sepsis
MeSH Terms: conditions — Sepsis | interventions — Interferon-gamma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interferon gamma-1b injection (Experimental): Patients randomized to the experimental arm will receive :
  Recombinant human interferon gamma-1b 2 X 106 IU, injectable solution. Subcutaneous injection every 24 hours for 3 consecutive days (3 total injections)
- Placebo injection (Placebo Comparator): Patients randomized to the placebo arm will receive saline injectable solution. Subcutaneous injection every 24 hours for 3 consecutive days (3 total injections)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Interferon Gamma 1-b — interferon gamma-1b 2 X 106 IU, injectable solution. Subcutaneous injection every 24 hours for 3 consecutive days (3 total injections)
Drug: Placebo — Patients randomized to the placebo arm will receive saline injectable solution. Subcutaneous injection every 24 hours for 3 consecutive days (3 total injections)
  Arms: Placebo injection

SUMMARY:
The vast majority of serious clinical situations leading to intensive care (septic shock, polytrauma, acute cerebral aggression, major surgery) are characterized by significant systemic inflammation. Recently, the existence of a common immune response pattern to acute aggression has been demonstrated, and with it the existence of a phenomenon known as post-aggressive immunosuppression (PAIS).

DETAILED DESCRIPTION:
The vast majority of serious clinical situations leading to intensive care (septic shock, polytrauma, acute cerebral aggression, major surgery) are characterized by significant systemic inflammation. Recently, the existence of a common immune response pattern to acute aggression has been demonstrated, and with it the existence of a phenomenon known as post-aggressive immunosuppression (PAIS).

This immunological adaptation, initially implemented as a host defense mechanism to protect against an overwhelming systemic reaction, can, if prolonged, lead to multiple complications resulting in significant delayed morbidity and mortality. Diagnosis is based on the use of immuno-inflammatory biomarkers, the most widely studied of which is monocyte expression of major histocompatibility complex type II molecules (mHLA-DR).

We have recently confirmed that PAIS can affect all types of patients admitted to the intensive care unit, but mainly occurs in the most severe patients. We also showed that the occurrence of PAIS was strongly associated with the subsequent occurrence of secondary infection and excess mortality.

Currently, there is no treatment with proven efficacy for PAIS, but several drugs have been shown to restore leukocyte function in-vitro. Several teams have reported the use of immunostimulatory molecules in patients with treatment failure, with a good safety profile and encouraging results. We believe that earlier treatment of patients with proven PAIS could improve their clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years old
* SOFA score for first 24 hours post-admission ≥ 6
* Mechanically ventilated at the time of inclusion (non-invasive ventilation (NIV) and high-flow nasal oxygen excluded)
* mHLA-DR< 8,000 AB/C measured between the 5th and 10th day after admission to the intensive care unit
* Patient affiliated to a social security scheme
* Written consent (relative/trusted person)

Exclusion Criteria:

* Patient with estimated life expectancy of less than 3 months
* Patients with a predicted remaining stay in intensive care < 72 hours
* Patient with pre-existing immunosuppression: solid cancer active or in remission for < 5 years, active hemopathy or in remission for < 5 years, systemic disease (including in the absence of specific treatment), solid organ transplant or marrow allograft patient, patient suffering from a HIV infection
* Patients with an expected prolonged duration of mechanical ventilation: comatose or vegetative patients (admission for severe stroke with Glasgow score < 8, patient resuscitated from an arterial stroke,) patients with tracheotomy for ENT problems, patients suffering from muscular disease (e.g. myopathy), patients on long-term mechanical ventilation
* Pregnant or breast-feeding women
* Contraindication of Imukin (hypersensitivity to interferon gamma-1b or known hypersensitivity to related products, such as another interferon)
* Patients on immunosuppressive therapy, including long-term corticosteroid therapy (>2.5mg/d prednisone equivalent)
* Patients with severe hepatic or renal insufficiency
* Patient included in another interventional clinical trial
* People under court protection and protected adults

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
number of days alive without mechanical ventilation | on Day 28 after drug administration
  number of days alive without mechanical ventilation on day 28 after randomization or on discharge from intensive care if this occurs before the 28th day

SECONDARY OUTCOMES:
Evaluate the efficacy of IFNy in correcting PAIS-defining biological abnormalities (re-ascension of mHLA-DR above 8,000 AB/C) between patients treated with recombinant interferon gamma 1-b versus placebo | Day 1 to Day 7 and at Day 28 post randomization
  Evolution of mHLA-DR measured at Day 0, Day 1, Day 2, Day 3, Day 7 and Day 28 or at discharge from intensive care if earlier (Day 0 corresponding to the day of inclusion in the study) between patients treated with recombinant interferon gamma 1-b versus placebo.
Evaluate, depending on the randomization arm, the kinetics of plasma inflammatory parameters between patients treated with recombinant interferon gamma 1-b versus placebo | Day 0, Day 3 and at Day 7 post randomization
  Evolution of inflammation markers (IL-1, IL-2, IL-6, IL-8, TNFa, etc.) measured in plasma at Day 0, Day 3 and Day 7, or at discharge from intensive care if it occurs before (Day 0 corresponding to the day of inclusion in the study) between patients treated with recombinant interferon gamma 1-b versus placebo
mortality at Day 28 and Day 90 after randomization | Day 28 and Day 90 after randomization
  Mortality rate at Day 28 and Day 90 after randomization between patients treated with recombinant interferon gamma 1-b versus placebo
incidence of nosocomial infections during intensive care unit stay | from Day 0 to Day 28 (or the discharge from intensive care)
  The incidence of nosocomial infections during an ICU stay between patients treated with recombinant interferon gamma 1-b versus placebo
number of days alive whithout antibiotic | Day 28 after drug administration
  Number of days alive without antibiotic assessed on day 28 after randomization between patients treated with recombinant interferon gamma 1-b versus placebo
length of stay in intensive care between patients | from Day 0 to Day 28 (or the discharge from intensive care)
  Number of days in intensive care between patients treated with recombinant interferon gamma 1-b versus placebo
- Compare organ failure score (SOFA) kinetics between patients treated with recombinant interferon gamma 1-b versus placebo | From inclusion to Day 7
  Kinetics of SOFA score assessed at inclusion and during the 7 days following inclusion between patients treated with recombinant interferon gamma 1-b versus placebo
Evaluate, depending on the randomization arm, the transcriptomic profile of circulating peripheral blood mononuclear cells count between patients treated with recombinant interferon gamma 1-b versus placebo | Day 0, Day 3 and Day 7 after randomization
  Evolution of the transcriptomic profile of circulating peripheral blood mononuclear cells (PBMCs) using scRNAseq analysis measured at Day 0, Day 3 and Day 7 or upon discharge from intensive care if this occurs earlier.
Evaluate, depending on the randomization arm the leucocyte count between patients treated with recombinant interferon gamma 1-b versus placebo | Day 0 to Day 7 and at Day 28 post randomization
  Evolution and kenetics of the leucocyte count measured at Day 0, Day 1, Day 2, Day 3, Day 7 and Day 28 or at discharge from intensive care if earlier (Day 0 corresponding to the day of inclusion in the study) between patients treated with recombinant interferon gamma 1-b versus placebo

CONTACTS AND LOCATIONS:
Overall Officials: Charles De ROQUETAILLADE, MD, Study Chair — APHP(ASSISTANCE PUBLIQUE DES HOPITAUX DE PARIS
Locations (2):
- France (2):
  - Dr de Roquetaillade, Paris
  - Pr Dépret, Paris

IPD SHARING:
Plan to Share IPD: Undecided